CLINICAL TRIAL: NCT05725824
Title: Novel Technology Adoption in the Audiology Clinic: Investigations of Ear Tip Performance, Perceptions, and Experiences
Brief Title: Investigations of Ear Tip Performance, Perceptions, and Experiences
Acronym: IETPPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002336
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Hearing Aids
Keywords: earmold; hearing aid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Third-party control (Active Comparator): Ear canal impressions will be will be packaged and sent to a professional third-party manufacturer for fabrication in an acrylic material-type. These will serve as the control earmolds, by which the in-house study/intervention earmolds will be compared against. To control for style of earmolds, all earmolds will be made in a skeleton style with a sound bore that accommodates size #13 tubing and a separate select-a-vent (SAV).
  Interventions: Device: BTE hearing aid with compatible earmolds
- In-house Study group_Resin (Experimental): Custom earmold impressions will be scanned and edited using computer-aided design software. These 3D earmold meshes will then be converted to g-code using licensed software and sent to a stereolithography 3D printer for fabrication. Participants will only wear these study earmolds for the duration of testing.To control for style of earmolds, all earmolds will be made in a skeleton style with a sound bore that accommodates size #13 tubing and a separate select-a-vent (SAV).
  Interventions: Device: BTE hearing aid with compatible earmolds
- In-house Study group_PLA (Experimental): Custom earmold impressions will be scanned and edited using computer-aided design software. These 3D earmold meshes will then be converted to g-code using licensed software and sent to a fused deposition modeling 3D printer for fabrication. Participants will only wear these study earmolds for the duration of testing. To control for style of earmolds, all earmolds will be made in a skeleton style with a sound bore that accommodates size #13 tubing and a separate select-a-vent (SAV).
  Interventions: Device: BTE hearing aid with compatible earmolds

INTERVENTIONS:
Device: BTE hearing aid with compatible earmolds — Hearing aids will be fit with three different types of customized earmolds. They will only wear each earmold group for the duration of the test (total = ~2.5 hours). Hearing aids will be programmed to a simulated mild, flat, sensorineural hearing loss of 30 dB HL from 250-8000Hz. A short washout period will follow completion of testing with ear earmold group.

SUMMARY:
Normal hearing participants will be fit with a hearing aid and different types of customized earmolds. Hearing aids will be programmed to a simulated mild, flat, sensorineural hearing loss of 30 dB HL from 250-8000Hz. Objective acoustic real ear measures and subjective ratings of sound quality and physical comfort will be evaluated and compared between earmolds. Findings will help researchers to better understand the impacts of different earmolds and how each might affect overall point-of-care.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing thresholds (<25 dB HL) at octave frequencies from 250-8000Hz.
* Normal otoscopy: patent ear canals with normal appearing eardrums and aerated middle ear, bilaterally.
* English as primary spoken language.

Exclusion Criteria:

* history of extensive or current outer or middle ear pathology.
* history of extensive outer or middle ear surgery.
* history of neurological or cognitive disorder.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 3rd Party Control, Then In-house PLA, Then In-house_RES: In this arm, participants were first fit and tested with a 3rd party control, then in-house PLA, then in-house_RES earmold
- In-house_RES, Then 3rd Party Control, Then In-house PLA: In this arm, participants were first fit and tested with a in-house_RES, then 3rd party control, then a in-house_PLA earmold
- In-house PLA, Then In-house_RES, Then 3rd Party Control: In this arm, participants were fit with a in-house PLA, then in-house_RES, then 3rd party control earmold.
Period: Overall Study
Arm/Group | 3rd Party Control, Then In-house PLA, Then In-house_RES | In-house_RES, Then 3rd Party Control, Then In-house PLA | In-house PLA, Then In-house_RES, Then 3rd Party Control
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Group: Crossover trial of 30 individuals with normal hearing
Arm/Group | Overall Group
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Black or African American | 2
  Hispanic/Latino | 7
  White/Non-hispanic | 14
  More than one race | 4

OUTCOME MEASURES:

1. Primary Outcome: Real Ear Measures
Description: Evaluation of ear canal acoustics with participant wearing a hearing aid and earmold type (3d party control, in-house_Resin, in-house_PLA). Then, a thin microphone tube is placed in the ear canal to measure the average amount gain (dB SPL) across various frequencies (250-8000Hz) while the participant sits in front of a speaker playing sound samples. Results are recorded in gain (dB SPL) across frequencies. Once complete, the earmold type is changed and recording is repeated until all ear mold material types have been tested for each individual. Arms/Groups were collapsed for RM-ANOVA to compare between various earmold types. A post-hoc paired t-test w/ Bonferroni correction was utilized to compare ear mold material types.
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: dB SPL
Groups:
- 3rd Party Control: Participants each wore and were tested with 3rd party control ear mold for 15 minutes.
- In-house_RES: Participants each wore and were tested with study in-house_RES ear mold for 15 minutes.
- In-house_PLA: Participants each wore and were tested with study in-house_PLA ear mold for 15 minutes.
Arm/Group | 3rd Party Control | In-house_RES | In-house_PLA
Number analyzed (Participants) | 30 | 30 | 30
dB SPL
  REAG_2000s | 61.23 (2.49) | 60.23 (2.01) | 60.5 (2.27)
  REAG_1000m | 64.53 (2.61) | 66.5 (2.73) | 66.23 (2.65)
  REAG_500l | 74.43 (2.01) | 75.4 (2.11) | 74.5 (2.00)
  REAG_1000l | 70.83 (2.57) | 72.23 (3.17) | 71.8 (3.40)
Statistical Analysis 1: Comparison: 3rd Party Control vs In-house_RES vs In-house_PLA; Test type: Superiority; p < 0.05, Repeated Measure Analysis of Variance

2. Primary Outcome: Outer Effectiveness of Auditory Rehabilitation (EAR) Questionnaire
Description: A questionnaire eliciting patient perception of physical comfort, quality of voice, and overall self-perceived satisfaction. Includes 12 items (5 point) that are scored on a 0 to 100, with 100 representing best possible function/rating
Time Frame: 2nd listening session appointment (15 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3rd Party Control | In-house_RES | In-house_PLA
Number analyzed (Participants) | 30 | 30 | 30
score on a scale
  PerceptVoice | 3.6 (0.97) | 3.77 (1.22) | 3.6 (1.22)
  NaturalSound | 3.17 (1.02) | 3.43 (1.25) | 3.3 (1.12)
  PhysComfort | 3.9 (0.97) | 4 (1.11) | 3.73 (1.05)
Statistical Analysis 1: Comparison: 3rd Party Control vs In-house_RES vs In-house_PLA; Test type: Superiority; p < 0.05, Repeated Measure Analysis of Variance

3. Primary Outcome: Physical Dimensions
Description: Physical dimensions of each ear mold type (3rd party Control, in-house_Resin, in-house_PLA) were taken using digital calipers in millimeters prior to being worn by participants.
Time Frame: Prior to 2nd listening session appointment (15 minutes)
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | 3rd Party Control | In-house_RES | In-house_PLA
Number analyzed (Participants) | 30 | 30 | 30
millimeters
  HeightTotal | 27.19 (2.01) | 27.73 (1.92) | 27.39 (1.85)
  WidthTotal | 21.42 (3.76) | 22.50 (3.55) | 22.23 (3.49)
  DepthTotal | 15.25 (1.66) | 13.88 (2.26) | 13.65 (1.86)
  Height_mEC | 7.72 (1.13) | 8.21 (0.91) | 8.38 (0.99)
  VentDiam | 2.56 (0.41) | 2.51 (0.37) | 2.23 (0.36)
Statistical Analysis 1: Comparison: 3rd Party Control vs In-house_RES vs In-house_PLA; Test type: Superiority; p < 0.05, Repeated Measure Analysis of Variance — Arms/Groups were collapsed for RM-ANOVA to compare between various earmold types. A post-hoc paired t-test w/ Bonferroni correction was utilized to compare ear mold material types

4. Primary Outcome: Production Variable
Description: The total raw cost ($) for each ear mold type (3rd party_control, in-house_RES, and in-house_PLA).
Time Frame: Prior to 2nd listening session appointment (15 minutes)
Measure: Mean (Standard Deviation); unit: dollars ($)
Arm/Group | 3rd Party Control | In-house_RES | In-house_PLA
Number analyzed (Participants) | 30 | 30 | 30
dollars ($) | 59.95 (0.00) | 1.29 (0.20) | 0.04 (0.00)
Statistical Analysis 1: Comparison: 3rd Party Control vs In-house_RES vs In-house_PLA; Test type: Superiority; p < 0.05, Repeated Measure Analysis of Variance

ADVERSE EVENTS:
Time Frame: 10-15 minutes brief wear time for each intervention earmold (3rd party_control, in-house_RES, in-house_PLA).
Description: Study involves minimal risk and limited wear time (15 minutes or less) and skin contact for each ear mold type. Participants were directly monitored while wearing the ear molds in the study. Participants did not keep or wear ear molds outside the study. Patients were not at risk of mortality or serious injury and were not monitored after their participation in the study.
Groups:
- 3rd Party Control, Then In-house_PLA, Then In-house_Resin: Each participant was fit with a 3rd party control, then in-house_PLA, then in-house_Resin ear mold. Each ear mold was worn for 10-15 minutes while outcome measures were collected. Each ear mold was separated by a brief washout period of 10 minutes.
  Study involves minimal risk and limited wear time (less than 15min) and skin contact for each earmold type. Participants were directly monitored during wear time. Patients are not at risk of mortality or serious injury.
- In-house_Resin, Then 3rd Party Control, Then In-house_PLA: Each participant was fit with a in-house_Resin, then 3rd party control, then in-house_PLA. Each ear mold was worn for 10-15 minutes while outcome measures were collected. Each ear mold was separated by a brief washout period of 10 minutes
  Study involves minimal risk and limited wear time (less than 15min) and skin contact for each earmold type. Participants were directly monitored during wear time. Patients are not at risk of mortality or serious injury.
- In-house_PLA, Then In-house_Resin, Then 3rd Party Control: Each participant was fit with a in-house_PLA, then in-house_Resin, then 3rd party control.Each ear mold was worn for 10-15 minutes while outcome measures were collected. Each ear mold was separated by a brief washout period of 10 minutes
  Study involves minimal risk and limited wear time (less than 15min) and skin contact for each earmold type. Participants were directly monitored during wear time. Patients are not at risk of mortality or serious injury.
Arm/Group | 3rd Party Control, Then In-house_PLA, Then In-house_Resin | In-house_Resin, Then 3rd Party Control, Then In-house_PLA | In-house_PLA, Then In-house_Resin, Then 3rd Party Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT05725824/Prot_SAP_000.pdf